CLINICAL TRIAL: NCT00605202
Title: Effect of Licorice and Hydrochlorothiazide on Plasma Potassium
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Professor Markku Savolainen, Oulu University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Lakritsi ja hypokalemia
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Results first posted 2009-12-09 (Estimated); Last update posted 2009-12-15 (Estimated); Status verified 2009-12

CONDITIONS: Hypokalemia
MeSH Terms: conditions — Hypokalemia | interventions — Hydrochlorothiazide; Glycyrrhiza glabra extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Licorice (Active Comparator)
  Interventions: Dietary Supplement: Licorice
- Licorice and HCTZ (Active Comparator)
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Hydrochlorothiazide — Hydrochlorothiazide 25 mg a day for 14 days.
  Other Names: Hydrex semi, ATC C03AA03
  Arms: Licorice and HCTZ
Dietary Supplement: Licorice — Licorice candy 32 grams a day for 14 days.
  Other Names: Pepe Original candy
  Arms: Licorice

SUMMARY:
This clinical trial is designed to study the effect of the combination of licorice and hydrochlorothiazide on plasma potassium levels in volunteers. In one arm, 10 healthy volunteers will be given 32 grams of licorice a day together with a 25 mg dose of daily hydrochlorothiazide for 14 days. This combination is compared with 32 grams of licorice a day for 14 days given in the other arm. The study is a randomized, open-label cross-over trial. There is at least a 3-week wash-out between the arms. The hypothesis is that the combination of licorice and hydrochlorothiazide will cause hypokalemia. The main outcome measure is the change in the plasma level of potassium between the arms.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer
* Age 18-40 years

Exclusion Criteria:

* Any continuous medication
* Any significant disease
* Hypotension or hypertension
* Allergy to licorice or hydrochlorothiazide
* Pregnancy and breast feeding
* Fear of needles and previous difficult blood samplings
* Substance abuse
* Participation in another clinical drug trial within 1 month of enrollment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Markku Savolainen, MD, Principal Investigator — Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Result] Hukkanen J, Ukkola O, Savolainen MJ. Effects of low-dose liquorice alone or in combination with hydrochlorothiazide on the plasma potassium in healthy volunteers. Blood Press. 2009;18(4):192-5. doi: 10.1080/08037050903072515. PMID 19562574

RESULTS

PARTICIPANT FLOW:
Groups:
- Licorice First, Then Licorice and HCTZ: Licorice 32 grams a day in the first intervention period, then licorice 32 grams a day together with Hydrochlorothiazide 25 mg once daily in the second intervention period.
- Licorice and HCTZ First, Then Licorice: Licorice 32 grams a day together with Hydrochlorothiazide 25 mg once daily in the first intervention period, then licorice 32 grams a day in the second intervention period.
Period: First Intervention
Arm/Group | Licorice First, Then Licorice and HCTZ | Licorice and HCTZ First, Then Licorice
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Washout Period of 3 Weeks
Arm/Group | Licorice First, Then Licorice and HCTZ | Licorice and HCTZ First, Then Licorice
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Licorice First, Then Licorice and HCTZ | Licorice and HCTZ First, Then Licorice
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  Finland | 10

OUTCOME MEASURES:

1. Primary Outcome: Plasma Potassium
Description: Plasma potassium measured with indirect ion specific electrode method
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Licorice | Licorice and HCTZ
Number analyzed (Participants) | 10 | 10
mmol/l
  Baseline | 4.0 (0.2) | 4.0 (0.3)
  2 weeks | 4.1 (0.3) | 3.7 (0.2)
Statistical Analysis 1: Comparison: Licorice vs Licorice and HCTZ; Statistical analysis applies to the change in the plasma potassium (baseline to 2 weeks) between arms; Test type: Superiority or Other; p = 0.007, t-test, 2 sided — P-value of the change in the plasma potassium (baseline to 2 weeks) between arms

ADVERSE EVENTS:
Groups:
- Licorice: Licorice 32 grams a day
- Licorice and HCTZ: Licorice 32 grams a day together with Hydrochlorothiazide 25 mg once daily
Arm/Group | Licorice | Licorice and HCTZ
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No